CLINICAL TRIAL: NCT03927300
Title: Telemonitoring Impact by the ApTelecare Software in Dialysis Patient
Acronym: MEDIA
Status: Completed | Type: Observational
Sponsor: Tmm Software (Industry)
Collaborators: Centre Hospitalier de Vichy (Other)
Responsible Party: Sponsor
Other Study IDs: KM-00153
Record Dates: First submitted 2019-04-12; First posted 2019-04-25 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Renal Failure; Dialysis Related Complication
Keywords: Home Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients without Telemonitoring with ApTelecare Software
- Patients with implementation of Telemonitoring with ApTelecare
  Interventions: Device: Telemonitoring Software

INTERVENTIONS:
Device: Telemonitoring Software — Recovery of retrospective data in dialysis patients follow or not follow by a telemonitoring application.
  Groups: Patients with implementation of Telemonitoring with ApTelecare

SUMMARY:
The investigators proposed to conduct a retrospective study to evaluate the impact of the implementation of apTeleCare software on the management of dialysis patients at home in terms of the number and duration of hospitalizations. For this purpose, the investigators will compare patients' data over a 2-year interval before the introduction of Telemonitoring (January 2012 and December 2013 inclusive - Group 1) with patients data who have benefited from this application (between August 2016 and July 2018).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) with no age limit;
* Patients receiving peritoneal dialysis on the investigation center between 2012 and 2014 (Group1) and between 2016 and 2018 (Group 2);
* Patient information in this retrospective study;

Exclusion Criteria:

* Patients who have started a peritoneal dialysis program before the periods of investigation;
* Patients who have been equipped with apTeleCare during the dialysis program;
* Subject under guardianship, curators or safeguard of justice;
* Patient not affiliated to a French social protection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a chronic renal failure who are take care in the dialysis unit. These patients are their peritoneal dialysis at home and use or not the telemonitoring software "ApTelecare".
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Cumulative duration (on retrospective two years of follow-up) of the unscheduled hospitalizations between the two patient groups. | up to two years.
Cumulative duration (on retrospective two years of follow-up) of the scheduled hospitalizations between the two patient groups. | up to two years.

SECONDARY OUTCOMES:
Total length of hospitalisation | For both groups. Every two months (follow-up visit) on a retrospective period of two years, the outcome 2 will be measured. The study duration will be of 5 months
Number of events of cardiovascular complications | For both groups. Every two months (follow-up visit) on a retrospective period of two years. The study duration will be of 5 months
Mortality rate | For both groups. At the end of this retrospective study (Study Period of 5 months).
Rate of peritoneal infections | For both groups. At the end of this retrospective study.(Study Period of 5 months).
Number of patient exit technique except death | For both groups. At the end of this retrospective study. (Study Period of 5 months).
  For example transplant, hemodialysis
Charlson score : Comorbidity index | baseline
  This scale measure the comorbidity symptoms of patients at the beginning of the care by the physician. The minimum score will be "0" and the maximum will be 39.
  Its validation is based on a prediction of health French insurance, as well as on several clinical areas such as oncology or nephrology.

CONTACTS AND LOCATIONS:
Locations (1):
- Matthieu Merlot, Montpellier, France